CLINICAL TRIAL: NCT01954966
Title: Multimodal Imaging of Progesterone/Neurosteroid Effects in Nicotine Addiction
Brief Title: Progesterone and Brain Imaging Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 811940; K24DA030301 (NIH)
Record Dates: First submitted 2012-11-06; First posted 2013-10-07 (Estimated); Results first posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Nicotine Dependence; Nicotine Withdrawal
Keywords: Nicotine; Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progesterone 200 mg capsules (Active Comparator): Subjects will be prescribed progesterone 200 mg capsules by the study Principal Investigator. Subjects will take 200 mg of progesterone daily for four days.
  Interventions: Drug: Progesterone
- Progesterone 200 mg look-alike capsules (Placebo Comparator): Subjects will be prescribed progesterone 200 mg look-alike placebo capsules by the study Principal Investigator. Subjects will take look-alike placebo capsules daily for four days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone — Participants will consume four pills of Progesterone over a period of four days. Participants will be asked to remain abstinent from smoking while taking Progesterone.
  Other Names: Prometrium
  Arms: Progesterone 200 mg capsules
Drug: Placebo — Participants will consume four pills of Placebo over a period of four days. Participants will be asked to remain abstinent from smoking while taking Placebo.
  Arms: Progesterone 200 mg look-alike capsules

SUMMARY:
Male and female smokers were recruited to undergo 2 phases of smoking cessation. Each phase was 4 days long and involved 3 brain-imaging scans, blood draws and an intervention involving progesterone or a matched placebo.

DETAILED DESCRIPTION:
The purpose of this study is to learn whether a sex hormone called progesterone is helpful in reducing cigarette smoking and craving for cigarettes. This study also includes brain imaging to measure possible effects of progesterone on certain neurochemicals. These neurochemicals are called gamma-aminobutyric acid (or GABA for short) and glutamate. Both nicotine and progesterone affect these brain chemicals.

Individuals wishing to participate in this study must be medically healthy men or women who smoke at least 10 cigarettes per day or greater. Participants must not suffer from a mental illness or use drugs other than nicotine and marijuana. Participants cannot have any implanted metallic devices such as pacemakers, orthodontic braces, or shrapnel. Participants must not have peanut allergies and must never have had a reaction to progesterone. Finally, participants cannot be taking any medications for anxiety, depression or insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Female and male smokers, aged 18 to 50 years;
* History of smoking greater than or equal to 10 cigarettes daily for the past year, as per self-report (periods of smoking abstinence within the last year will be exclusionary at PI discretion);
* Not seeking treatment at the time of the study for nicotine dependence;
* Have a Fagerstrom Test for Nicotine Dependence (FTND) score of at least 3 and a Carbon Monoxide (CO) level greater than or equal to 11 ppm;
* Clean urine drug screen (marijuana is permissible);
* In good health as verified by medical history;
* For women, not pregnant as determined by pregnancy screening, nor breast feeding.

Exclusion Criteria:

* History of major medical illness: including liver diseases, abnormal vaginal bleeding, suspected or known malignancy; thrombophlebitis; deep vein thrombosis; pulmonary embolus; clotting or bleeding disorders; heart disease; diabetes; history of stroke or other medical conditions that the physician investigator deems as contraindicated for the patient to be in the study;
* Regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics) and recent (within previous year) psychiatric diagnosis and treatment for Axis I disorders including major depression, bipolar affective disorder, generalized anxiety disorder, post-traumatic stress disorder and panic disorder;
* Lifetime history of schizophrenia or other psychotic disorder;
* Lifetime substance dependence disorder, excepting nicotine, alcohol and marijuana, as per SCID interview
* Substance use disorders within the previous 2 years, excepting nicotine, as per SCID interview
* Regular use of any other tobacco products than cigarettes, including smokeless tobacco and nicotine products;
* Known allergy to progesterone or peanuts (vehicle for micronized progesterone).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia N Epperson, M.D., Principal Investigator — Associate Professor of Psychiatry, University of Pennsylvania
Locations (1):
- Penn Center for Women's Behavioral Wellness, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Epperson CN, O'Malley S, Czarkowski KA, Gueorguieva R, Jatlow P, Sanacora G, Rothman DL, Krystal JH, Mason GF. Sex, GABA, and nicotine: the impact of smoking on cortical GABA levels across the menstrual cycle as measured with proton magnetic resonance spectroscopy. Biol Psychiatry. 2005 Jan 1;57(1):44-8. doi: 10.1016/j.biopsych.2004.09.021. PMID 15607299
- [Background] Cai K, Nanga RP, Lamprou L, Schinstine C, Elliott M, Hariharan H, Reddy R, Epperson CN. The impact of gabapentin administration on brain GABA and glutamate concentrations: a 7T (1)H-MRS study. Neuropsychopharmacology. 2012 Dec;37(13):2764-71. doi: 10.1038/npp.2012.142. Epub 2012 Aug 8. PMID 22871916
- [Background] Epperson CN, Toll B, Wu R, Amin Z, Czarkowski KA, Jatlow P, Mazure CM, O'Malley SS. Exploring the impact of gender and reproductive status on outcomes in a randomized clinical trial of naltrexone augmentation of nicotine patch. Drug Alcohol Depend. 2010 Nov 1;112(1-2):1-8. doi: 10.1016/j.drugalcdep.2010.04.021. Epub 2010 Jun 19. PMID 20561758
- [Background] Mason GF, Petrakis IL, de Graaf RA, Gueorguieva R, Guidone E, Coric V, Epperson CN, Rothman DL, Krystal JH. Cortical gamma-aminobutyric acid levels and the recovery from ethanol dependence: preliminary evidence of modification by cigarette smoking. Biol Psychiatry. 2006 Jan 1;59(1):85-93. doi: 10.1016/j.biopsych.2005.06.009. Epub 2005 Nov 14. PMID 16289397
- [Background] Cosgrove KP, Mitsis EM, Bois F, Frohlich E, Tamagnan GD, Krantzler E, Perry E, Maciejewski PK, Epperson CN, Allen S, O'malley S, Mazure CM, Seibyl JP, van Dyck CH, Staley JK. 123I-5-IA-85380 SPECT imaging of nicotinic acetylcholine receptor availability in nonsmokers: effects of sex and menstrual phase. J Nucl Med. 2007 Oct;48(10):1633-40. doi: 10.2967/jnumed.107.042317. Epub 2007 Sep 14. PMID 17873128
- [Derived] Novick AM, Duffy KA, Johnson RL, Sammel MD, Cao W, Strasser AA, Sofuoglu M, Kuzma A, Loughead J, Morrow AL, Epperson CN. Effect of progesterone administration in male and female smokers on nicotine withdrawal and neural response to smoking cues: role of progesterone conversion to allopregnanolone. Biol Sex Differ. 2022 Oct 23;13(1):60. doi: 10.1186/s13293-022-00472-w. PMID 36274158
- [Derived] Novick AM, Duffy KA, Johnson RL, Sammel MD, Cao W, Strasser AA, Sofuoglu M, Kuzma A, Loughead J, Epperson CN. Progesterone Increases Nicotine Withdrawal and Anxiety in Male but Not Female Smokers During Brief Abstinence. Nicotine Tob Res. 2022 Nov 12;24(12):1898-1905. doi: 10.1093/ntr/ntac146. PMID 35713950
- See also: Center Website — http://www.med.upenn.edu/womenswellness/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 81 participants who were enrolled in the study, but N = 15 were lost to early follow-up before they could be randomized. Therefore, only N = 66 participants were randomized (N = 34 randomized to receive placebo first, N = 32 randomized to receive progesterone first).
Groups:
- Placebo First, Progesterone Second: This group was randomized to receive placebo during phase 1 of the crossover trial and progesterone during phase 2 of the crossover trial.
- Progesterone First, Placebo Second: This group was randomized to receive progesterone during phase 1 of the crossover trial and placebo during phase 2 of the crossover trial.
Period: Overall Study
Arm/Group | Placebo First, Progesterone Second | Progesterone First, Placebo Second
Started | 34 | 32
Completed Week 1 of Intervention (Drug Assigned to Receive First) | 30 | 30
Started Phase 2 After Washout Period (1-2 Week for Males, 1-3 Month for Females) | 30 | 30
Completed Week 2 of Intervention (Drug Assigned to Receive Second) | 24 | 28
Completed | 24 | 28
Not Completed | 10 | 4

BASELINE CHARACTERISTICS:
Population: A total of 81 participants were enrolled, but N = 15 were lost to early follow-up and were not randomized. Therefore, the analysis cohort includes N = 66 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First, Progesterone Second | Progesterone First, Placebo Second | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: N = 1 participant was missing age information in the progesterone first, placebo second randomization group.
  years
    number analyzed (Participants) | 34 | 31 | 65
    (all) | 35.5 (9.0) | 37.7 (7.6) | 36.6 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 18 | 15 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 31 | 27 | 58
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 22 | 44
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: GABA Pre and Post Progesterone Administration (Dorsal Anterior Cingulate Cortex [DACC])
Description: GABA concentrations (collected in the Dorsal Anterior Cingulate Cortex [DACC]) will be obtained using the non-invasive neuroimaging method of proton magnetic resonance spectroscopy (1H-MRS) both before and after placebo administration and smoking abstinence. In total subjects will undergo 6 1H-MRS scans. The 6 1H-MRS scans take place over a period of approximately 1-2 months. Each paradigm (placebo/progesterone) takes approximately one week, with an approximately two-week wash in between paradigms for men and an approximately 1-month wash in between paradigms for women. The subject will undergo a smoking session on Test Day #1 and Test Day #5, MRS scans are conducted on Test Day #2 (2 scans) and Test Day #5 (1 scan).
  Minimal data is available for the primary outcome due to substantial issues with the 7T scanner. All subsequent scans were conducted on a 3T scanner which does not have the capacity to collect data on GABA.
Time Frame: Test Day #2 and Test Day #5 - 6 total scans over the period of 2-3 months.
Population: Some values were missing due to visits for these individuals scheduled after there were issues with the 7T scanner, so data could not be collected for other participants.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 10 | 12
mg/dl
  Test day 2 (baseline, pre-scan) | 1.23 (0.05) | 1.17 (0.04)
  Test day 2 (post-scan): number analyzed (Participants) | 10 | 11
  Test day 2 (post-scan) | 1.28 (0.05) | 1.24 (0.04)
  Test day 5 (pre-smoking): number analyzed (Participants) | 10 | 10
  Test day 5 (pre-smoking) | 1.21 (0.05) | 1.17 (0.05)

2. Primary Outcome: GABA Pre and Post Progesterone Administration (Dorsolateral Pre-Frontal Cortex [DLPFC])
Description: GABA concentrations (collected in the Dorsolateral Pre-Frontal Cortex [DLPFC]) will be obtained using the non-invasive neuroimaging method of proton magnetic resonance spectroscopy (1H-MRS) both before and after placebo administration and smoking abstinence. In total subjects will undergo 6 1H-MRS scans. The 6 1H-MRS scans take place over a period of approximately 1-2 months. Each paradigm (placebo/progesterone) takes approximately one week, with an approximately two-week wash in between paradigms for men and an approximately 1-month wash in between paradigms for women. The subject will undergo a smoking session on Test Day #1 and Test Day #5, MRS scans are conducted on Test Day #2 (2 scans) and Test Day #5 (1 scan).
  Minimal data is available for the primary outcome due to substantial issues with the 7T scanner. All subsequent scans were conducted on a 3T scanner which does not have the capacity to collect data on GABA.
Time Frame: Test Day #2 and Test Day #5 - 6 total scans over the period of 2-3 months.
Population: Some data was not collected for participants due to issues with the 7T.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 10 | 12
mg/dl
  Day 2- pre scan | 1.18 (0.13) | 1.20 (0.11)
  Day 2- post scan: number analyzed (Participants) | 10 | 11
  Day 2- post scan | 1.05 (0.13) | 0.98 (0.12)
  Day 5- after scan, pre smoking | 1.06 (0.11) | 1.11 (0.16)

3. Secondary Outcome: Symptoms During Nicotine Abstinence (NWSC)
Description: Withdrawal symptoms will be measured using the Nicotine Withdrawal Symptoms Checklist (NWSC). The scale ranges from a minimum of 0 to a maximum of 28, with higher scores indicating greater withdrawal (more withdrawal symptoms, higher intensity/severity of withdrawal).
Time Frame: Day 1 (pre and post smoking session, day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some secondary outcome data is missing because missed visits and dropouts occurred due to the number of visits required for the study. The study team attempted to limit missing data with payment at each visit for contingency management and allowing participants to continue in the study if individual visits were missed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Nicotine withdrawal symptoms checklist (NWSC); day 1 pre 1st smoking session: number analyzed (Participants) | 58 | 61
  Nicotine withdrawal symptoms checklist (NWSC); day 1 pre 1st smoking session | 6.00 (0.59) | 6.15 (0.58)
  Nicotine withdrawal symptoms checklist (NWSC); day 1 post 1st smoking session: number analyzed (Participants) | 56 | 59
  Nicotine withdrawal symptoms checklist (NWSC); day 1 post 1st smoking session | 4.84 (0.60) | 4.48 (0.59)
  Nicotine withdrawal symptoms checklist (NWSC); day 2 pre-scan: number analyzed (Participants) | 59 | 60
  Nicotine withdrawal symptoms checklist (NWSC); day 2 pre-scan | 5.67 (0.59) | 4.92 (0.59)
  Nicotine withdrawal symptoms checklist (NWSC); day 2 post-scan | 5.37 (0.60) | 5.25 (0.60)
  Nicotine withdrawal symptoms checklist (NWSC); day 3 abstinence AM: number analyzed (Participants) | 55 | 55
  Nicotine withdrawal symptoms checklist (NWSC); day 3 abstinence AM | 7.07 (0.60) | 7.62 (0.60)
  Nicotine withdrawal symptoms checklist (NWSC); day 3 abstinence PM: number analyzed (Participants) | 56 | 56
  Nicotine withdrawal symptoms checklist (NWSC); day 3 abstinence PM | 6.99 (0.60) | 7.88 (0.60)
  Nicotine withdrawal symptoms checklist (NWSC); day 4 abstinence AM: number analyzed (Participants) | 55 | 55
  Nicotine withdrawal symptoms checklist (NWSC); day 4 abstinence AM | 7.33 (0.60) | 7.66 (0.60)
  Nicotine withdrawal symptoms checklist (NWSC); day 4 abstinence PM: number analyzed (Participants) | 54 | 53
  Nicotine withdrawal symptoms checklist (NWSC); day 4 abstinence PM | 7.19 (0.60) | 7.32 (0.61)
  Nicotine withdrawal symptoms checklist (NWSC); day 5 pre-smoking: number analyzed (Participants) | 55 | 50
  Nicotine withdrawal symptoms checklist (NWSC); day 5 pre-smoking | 7.01 (0.60) | 7.34 (0.62)
  Nicotine withdrawal symptoms checklist (NWSC); day 5 post-smoking: number analyzed (Participants) | 54 | 44
  Nicotine withdrawal symptoms checklist (NWSC); day 5 post-smoking | 4.60 (0.60) | 4.82 (0.65)

4. Secondary Outcome: Brief Questionnaire on Smoking Urges (BQSU)
Description: Craving will be assessed using the Brief Questionnaire on Smoking Urges (BQSU). It ranges from 7-70 with higher levels indicating higher levels of nicotine craving.
Time Frame: as for outcome 3
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 1; pre-1st smoking session: number analyzed (Participants) | 51 | 56
  Day 1; pre-1st smoking session | 40.89 (2.23) | 41.94 (2.16)
  Day 1; post-1st smoking session: number analyzed (Participants) | 45 | 52
  Day 1; post-1st smoking session | 30.45 (2.33) | 25.77 (2.22)
  Day 2; pre-1st scan: number analyzed (Participants) | 48 | 54
  Day 2; pre-1st scan | 38.47 (2.28) | 34.34 (2.19)
  Day 2; post-2nd scan: number analyzed (Participants) | 46 | 49
  Day 2; post-2nd scan | 38.81 (2.31) | 37.98 (2.26)
  Day 3; abstinence AM: number analyzed (Participants) | 48 | 49
  Day 3; abstinence AM | 41.91 (2.28) | 41.82 (2.26)
  Day 3; abstinence PM: number analyzed (Participants) | 48 | 50
  Day 3; abstinence PM | 40.84 (2.28) | 42.03 (2.25)
  Day 4; abstinence AM: number analyzed (Participants) | 47 | 49
  Day 4; abstinence AM | 40.90 (2.30) | 40.29 (2.26)
  Day 4; abstinence PM: number analyzed (Participants) | 48 | 47
  Day 4; abstinence PM | 39.23 (2.28) | 37.68 (2.30)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 49 | 44
  Day 5; after scan, pre-smoking | 41.95 (2.26) | 42.38 (2.35)
  Day 5; after smoking: number analyzed (Participants) | 47 | 40
  Day 5; after smoking | 27.64 (2.29) | 28.22 (2.42)

5. Secondary Outcome: Tiffany Questionnaire on Smoking Urges (TQSU)
Description: Craving will also be assessed using the Tiffany Questionnaire for Smoking Urges. It ranges from 32 to 224 with higher scores indicated higher levels of smoking urges/craving.
Time Frame: Day 1 (pre smoking session, day 3 (PM), day 4 (PM), day 5 (pre smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 1; pre-1st smoking session: number analyzed (Participants) | 55 | 60
  Day 1; pre-1st smoking session | 143.45 (5.13) | 140.31 (5.00)
  Day 3; abstinence PM: number analyzed (Participants) | 52 | 50
  Day 3; abstinence PM | 138.46 (5.23) | 140.77 (5.29)
  Day 4; abstinence PM: number analyzed (Participants) | 54 | 48
  Day 4; abstinence PM | 139.11 (5.17) | 135.88 (5.36)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 56 | 48
  Day 5; after scan, pre-smoking | 146.22 (5.11) | 141.08 (5.36)

6. Secondary Outcome: Profile of Mood States (POMS) Subscale: Tension-Anxiety
Description: Profile of Mood States (POMS) Subscale: Tension-Anxiety. This subscale ranges from 0-28 with higher levels indicating greater tension/anxiety.
Time Frame: Day 2 (pre and post scan), Day 5 (pre smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 57 | 59
  Day 2; pre-1st scan | 2.88 (0.46) | 2.57 (0.46)
  Day 2; post- 2nd scan: number analyzed (Participants) | 55 | 56
  Day 2; post- 2nd scan | 3.55 (0.47) | 3.11 (0.47)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 55 | 48
  Day 5; after scan, pre-smoking | 4.85 (0.47) | 3.70 (0.50)

7. Secondary Outcome: Profile of Mood States (POMS) Subscale: Depression-Dejection
Description: Profile of Mood States (POMS) Subscale: Depression-Dejection. This subscale ranges from 0-60 with higher levels indicating greater depression/dejection.
Time Frame: Day 2 (pre and post scan), Day 5 (pre smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 59
  Day 2; pre-1st scan | 1.09 (0.34) | 0.64 (0.34)
  Day 2; post-2nd scan: number analyzed (Participants) | 55 | 56
  Day 2; post-2nd scan | 1.30 (0.35) | 0.88 (0.35)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 55 | 48
  Day 5; after scan, pre-smoking | 1.66 (0.35) | 1.81 (0.37)

8. Secondary Outcome: Profile of Mood States (POMS) Subscale: Anger-Hostility
Description: Profile of Mood States (POMS) Subscale: Anger-Hostility. This scale ranges from 0 to 48 with higher levels indicating higher levels of anger/hostility.
Time Frame: Day 2 (pre and post scan), Day 5 (pre smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 59
  Day 2; pre-1st scan | 0.94 (0.36) | 0.83 (0.36)
  Day 2; post-2nd scan: number analyzed (Participants) | 55 | 56
  Day 2; post-2nd scan | 1.55 (0.37) | 1.41 (0.37)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 55 | 48
  Day 5; after scan, pre-smoking | 2.70 (0.37) | 2.36 (0.39)

9. Secondary Outcome: Profile of Mood States (POMS) Subscale: Fatigue
Description: Profile of Mood States (POMS) Subscale: Fatigue. This subscale ranges from 0 to 28 with higher scores indicating higher levels of fatigue.
Time Frame: Day 2 (pre and post scan), Day 5 (pre smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 58
  Day 2; pre-1st scan | 2.17 (0.48) | 1.77 (0.49)
  Day 2; post-2nd scan: number analyzed (Participants) | 54 | 56
  Day 2; post-2nd scan | 2.84 (0.50) | 3.63 (0.49)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 55 | 47
  Day 5; after scan, pre-smoking | 3.66 (0.50) | 3.10 (0.53)

10. Secondary Outcome: Profile of Mood State (POMS) Subscale: Vigor
Description: Profile of Mood State (POMS) Subscale: Vigor. Subscale ranges from 0 to 32, with higher levels indicating higher levels of vigor.
Time Frame: Day 2 (pre and post scan), Day 5 (pre smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 58 | 56
  Day 2; pre-1st scan | 18.71 (0.94) | 18.71 (0.95)
  Day 2; post-2nd scan: number analyzed (Participants) | 54 | 53
  Day 2; post-2nd scan | 16.74 (0.96) | 16.73 (0.96)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 54 | 47
  Day 5; after scan, pre-smoking | 16.71 (0.96) | 16.39 (0.98)

11. Secondary Outcome: Profile of Mood States (POMS) Subscale: Confusion-Bewilderment
Description: Profile of Mood States (POMS) Subscale: Confusion-Bewilderment. Ranges from 0 to 28 with higher levels indicating higher levels of confusion/bewilderment.
Time Frame: Day 2 (pre and post scan), Day 5 (pre smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 59
  Day 2; pre-1st scan | 2.47 (0.35) | 2.31 (0.35)
  Day 2; post-2nd scan: number analyzed (Participants) | 55 | 56
  Day 2; post-2nd scan | 2.95 (0.36) | 2.98 (0.35)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 55 | 48
  Day 5; after scan, pre-smoking | 3.46 (0.36) | 2.80 (0.37)

12. Secondary Outcome: Visual Analog Scale (VAS) Question: Headache
Description: Visual Analog Scale (VAS) question: Headache. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 6.50 (2.55) | 7.59 (2.54)
  Day 2; post-2nd scan: number analyzed (Participants) | 59 | 58
  Day 2; post-2nd scan | 5.74 (2.55) | 9.39 (2.57)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 9.15 (2.65) | 14.71 (2.65)
  Day 3; abstinence PM: number analyzed (Participants) | 53 | 54
  Day 3; abstinence PM | 8.86 (2.67) | 10.93 (2.65)
  Day 4; abstinence AM: number analyzed (Participants) | 54 | 53
  Day 4; abstinence AM | 10.88 (2.65) | 7.70 (2.67)
  Day 4; abstinence PM: number analyzed (Participants) | 54 | 51
  Day 4; abstinence PM | 11.83 (2.65) | 12.78 (2.71)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 9.05 (2.59) | 13.36 (2.71)
  Day 5; after smoking: number analyzed (Participants) | 49 | 57
  Day 5; after smoking | 11.93 (2.59) | 11.67 (2.75)

13. Secondary Outcome: Visual Analog Scale (VAS) Question: Hunger
Description: Visual Analog Scale (VAS) question: Hunger. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 34.60 (3.73) | 40.23 (3.70)
  Day 2; post-2nd scan: number analyzed (Participants) | 59 | 58
  Day 2; post-2nd scan | 28.63 (3.75) | 22.20 (3.73)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 24.88 (3.85) | 33.40 (3.85)
  Day 3; abstinence PM: number analyzed (Participants) | 54 | 53
  Day 3; abstinence PM | 27.72 (3.87) | 31.95 (3.85)
  Day 4; abstinence AM: number analyzed (Participants) | 54 | 53
  Day 4; abstinence AM | 27.94 (3.85) | 34.64 (3.88)
  Day 4; abstinence PM: number analyzed (Participants) | 54 | 51
  Day 4; abstinence PM | 25.57 (3.85) | 29.27 (3.93)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 28.22 (3.78) | 35.22 (3.93)
  Day 5; after smoking: number analyzed (Participants) | 57 | 49
  Day 5; after smoking | 28.63 (3.78) | 32.61 (3.99)

14. Secondary Outcome: Visual Analog Scale (VAS) Question: Nauseous
Description: Visual Analog Scale (VAS) question: Nauseous. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 58 | 59
  Day 2; pre-1st scan | 5.52 (2.07) | 4.92 (2.06)
  Day 2; post-2nd scan: number analyzed (Participants) | 54 | 59
  Day 2; post-2nd scan | 6.31 (2.07) | 5.43 (2.08)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 6.01 (2.14) | 10.44 (2.14)
  Day 3; abstinence PM: number analyzed (Participants) | 53 | 53
  Day 3; abstinence PM | 8.07 (2.15) | 9.85 (2.14)
  Day 4; abstinence AM: number analyzed (Participants) | 51 | 54
  Day 4; abstinence AM | 6.07 (2.14) | 8.22 (2.15)
  Day 4; abstinence PM: number analyzed (Participants) | 51 | 54
  Day 4; abstinence PM | 6.60 (2.18) | 10.29 (2.18)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 6.51 (2.10) | 10.34 (2.18)
  Day 5; after smoking: number analyzed (Participants) | 57 | 49
  Day 5; after smoking | 8.00 (2.10) | 11.41 (2.22)

15. Secondary Outcome: Visual Analog Scale (VAS) Question: Heartburn.
Description: Visual Analog Scale (VAS) question: Heartburn. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 3.11 (1.70) | 2.35 (1.69)
  Day 2; post-2nd scan: number analyzed (Participants) | 59 | 58
  Day 2; post-2nd scan | 4.30 (1.70) | 4.06 (1.71)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 5.46 (1.76) | 3.27 (1.76)
  Day 3; abstinence PM: number analyzed (Participants) | 53 | 54
  Day 3; abstinence PM | 6.00 (1.78) | 4.55 (1.76)
  Day 4; abstinence AM: number analyzed (Participants) | 54 | 53
  Day 4; abstinence AM | 7.31 (1.76) | 6.50 (1.78)
  Day 4; abstinence PM: number analyzed (Participants) | 51 | 54
  Day 4; abstinence PM | 5.51 (1.76) | 5.56 (1.80)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 4.33 (1.73) | 5.30 (1.80)
  Day 5; after smoking: number analyzed (Participants) | 57 | 49
  Day 5; after smoking | 4.56 (1.73) | 6.37 (1.83)

16. Secondary Outcome: Visual Analog Scale (VAS) Question: Tired
Description: Visual Analog Scale (VAS) question: Tired. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 24.15 (3.76) | 18.62 (3.74)
  Day 2; post-2nd scan: number analyzed (Participants) | 59 | 58
  Day 2; post-2nd scan | 29.67 (3.76) | 40.92 (3.79)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 21.64 (3.89) | 27.24 (3.89)
  Day 3; abstinence PM: number analyzed (Participants) | 53 | 54
  Day 3; abstinence PM | 30.82 (3.91) | 35.53 (3.89)
  Day 4; abstinence AM: number analyzed (Participants) | 54 | 53
  Day 4; abstinence AM | 31.73 (3.89) | 27.99 (3.92)
  Day 4; abstinence PM: number analyzed (Participants) | 54 | 51
  Day 4; abstinence PM | 30.69 (3.89) | 28.51 (3.97)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 33.94 (3.82) | 32.06 (3.97)
  Day 5; after smoking: number analyzed (Participants) | 57 | 49
  Day 5; after smoking | 31.22 (3.82) | 34.79 (4.03)

17. Secondary Outcome: Visual Analog Scale (VAS) Question: Irritable
Description: Visual Analog Scale (VAS) question: Irritable. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 7.50 (3.42) | 5.71 (3.40)
  Day 2; post-2nd scan: number analyzed (Participants) | 59 | 58
  Day 2; post-2nd scan | 13.20 (3.42) | 13.01 (3.44)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 24.80 (3.54) | 24.56 (3.54)
  Day 3; abstinence PM: number analyzed (Participants) | 53 | 54
  Day 3; abstinence PM | 23.97 (3.56) | 25.49 (3.54)
  Day 4; abstinence AM: number analyzed (Participants) | 54 | 53
  Day 4; abstinence AM | 30.79 (3.54) | 29.58 (3.56)
  Day 4; abstinence PM: number analyzed (Participants) | 51 | 54
  Day 4; abstinence PM | 26.50 (3.54) | 30.11 (3.61)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 23.23 (3.47) | 22.96 (3.61)
  Day 5; after smoking: number analyzed (Participants) | 57 | 49
  Day 5; after smoking | 13.45 (3.47) | 15.52 (3.66)

18. Secondary Outcome: Visual Analog Scale (VAS) Question: Energetic
Description: Visual Analog Scale (VAS) question: Energetic. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 54.86 (3.68) | 67.01 (3.66)
  Day 2; post-2nd scan: number analyzed (Participants) | 59 | 58
  Day 2; post-2nd scan | 55.18 (3.68) | 21.03 (3.69)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 56.14 (3.77) | 58.11 (3.77)
  Day 3; abstinence PM: number analyzed (Participants) | 53 | 54
  Day 3; abstinence PM | 56.13 (3.79) | 50.12 (3.77)
  Day 4; abstinence AM: number analyzed (Participants) | 54 | 53
  Day 4; abstinence AM | 55.62 (3.77) | 54.89 (3.79)
  Day 4; abstinence PM: number analyzed (Participants) | 54 | 51
  Day 4; abstinence PM | 53.45 (3.77) | 56.77 (3.83)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 51.47 (3.72) | 56.64 (3.83)
  Day 5; after smoking: number analyzed (Participants) | 57 | 49
  Day 5; after smoking | 54.79 (3.72) | 54.70 (3.87)

19. Secondary Outcome: Visual Analog Scale (VAS) Question: Relaxed
Description: Visual Analog Scale (VAS) question: Relaxed. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 58 | 58
  Day 2; pre-1st scan | 72.66 (3.64) | 73.87 (3.64)
  Day 2; post-2nd scan: number analyzed (Participants) | 56 | 58
  Day 2; post-2nd scan | 67.77 (3.64) | 63.65 (3.67)
  Day 3; abstinence AM: number analyzed (Participants) | 53 | 52
  Day 3; abstinence AM | 63.87 (3.75) | 55.85 (3.77)
  Day 3; abstinence PM: number analyzed (Participants) | 52 | 52
  Day 3; abstinence PM | 57.69 (3.77) | 54.08 (3.77)
  Day 4; abstinence AM: number analyzed (Participants) | 53 | 51
  Day 4; abstinence AM | 57.83 (3.75) | 55.37 (3.79)
  Day 4; abstinence PM: number analyzed (Participants) | 53 | 49
  Day 4; abstinence PM | 63.46 (3.75) | 63.45 (3.84)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 56 | 50
  Day 5; after scan, pre-smoking | 62.45 (3.68) | 67.65 (3.81)
  Day 5; after smoking: number analyzed (Participants) | 56 | 48
  Day 5; after smoking | 67.99 (3.86) | 67.55 (3.68)

20. Secondary Outcome: Visual Analog Scale (VAS) Question: Talkative
Description: as for outcome 12
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 54.17 (3.76) | 57.46 (3.75)
  Day 2; post-2nd scan: number analyzed (Participants) | 59 | 58
  Day 2; post-2nd scan | 50.61 (3.76) | 51.46 (3.78)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 51.43 (3.84) | 50.34 (3.84)
  Day 3; abstinence PM: number analyzed (Participants) | 53 | 54
  Day 3; abstinence PM | 48.14 (3.86) | 47.04 (3.84)
  Day 4; abstinence AM: number analyzed (Participants) | 54 | 53
  Day 4; abstinence AM | 49.67 (3.84) | 50.71 (3.86)
  Day 4; abstinence PM: number analyzed (Participants) | 54 | 51
  Day 4; abstinence PM | 50.48 (3.84) | 49.27 (3.90)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 52.74 (3.80) | 56.19 (3.90)
  Day 5; after smoking: number analyzed (Participants) | 57 | 49
  Day 5; after smoking | 54.26 (3.80) | 53.12 (3.93)

21. Secondary Outcome: Visual Analog Scale (VAS) Question: Happy
Description: Visual Analog Scale (VAS) question: Happy. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 76.62 (3.39) | 79.70 (3.37)
  Day 2; post-2nd scan: number analyzed (Participants) | 59 | 58
  Day 2; post-2nd scan | 70.98 (3.39) | 71.34 (3.40)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 66.22 (3.47) | 64.04 (3.47)
  Day 3; abstinence PM: number analyzed (Participants) | 53 | 54
  Day 3; abstinence PM | 65.10 (3.49) | 61.30 (3.47)
  Day 4; abstinence AM: number analyzed (Participants) | 54 | 53
  Day 4; abstinence AM | 62.76 (3.47) | 60.58 (3.49)
  Day 4; abstinence PM: number analyzed (Participants) | 54 | 51
  Day 4; abstinence PM | 61.99 (3.47) | 63.95 (3.52)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 66.59 (3.42) | 63.46 (3.52)
  Day 5; after smoking: number analyzed (Participants) | 57 | 49
  Day 5; after smoking | 70.07 (3.42) | 67.87 (3.56)

22. Secondary Outcome: Visual Analog Scale (VAS) Question: Nervous
Description: Visual Analog Scale (VAS) question: Nervous. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 13.24 (2.50) | 10.26 (2.49)
  Day 2; post-2nd scan: number analyzed (Participants) | 59 | 58
  Day 2; post-2nd scan | 10.91 (2.50) | 8.46 (2.52)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 7.19 (2.57) | 8.22 (2.57)
  Day 3; abstinence PM: number analyzed (Participants) | 53 | 54
  Day 3; abstinence PM | 9.56 (2.59) | 9.24 (2.57)
  Day 4; abstinence AM: number analyzed (Participants) | 54 | 53
  Day 4; abstinence AM | 9.36 (2.57) | 11.37 (2.59)
  Day 4; abstinence PM: number analyzed (Participants) | 54 | 51
  Day 4; abstinence PM | 10.83 (2.57) | 10.66 (2.62)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 10.79 (2.53) | 12.15 (2.62)
  Day 5; after smoking: number analyzed (Participants) | 57 | 49
  Day 5; after smoking | 7.64 (2.53) | 11.94 (2.65)

23. Secondary Outcome: Visual Analog Scale (VAS) Question: Sad
Description: Visual Analog Scale (VAS) question: Sad. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 3.95 (1.87) | 2.09 (1.85)
  Day 2; post-2nd scan: number analyzed (Participants) | 59 | 58
  Day 2; post-2nd scan | 6.77 (1.87) | 4.48 (1.88)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 5.67 (1.93) | 10.51 (1.93)
  Day 3; abstinence PM: number analyzed (Participants) | 53 | 54
  Day 3; abstinence PM | 4.36 (1.95) | 9.07 (1.93)
  Day 4; abstinence AM: number analyzed (Participants) | 54 | 53
  Day 4; abstinence AM | 8.54 (1.93) | 8.47 (1.95)
  Day 4; abstinence PM: number analyzed (Participants) | 54 | 51
  Day 4; abstinence PM | 7.32 (1.93) | 8.65 (1.98)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 3.87 (1.89) | 12.47 (1.98)
  Day 5; after smoking: number analyzed (Participants) | 57 | 49
  Day 5; after smoking | 2.95 (1.89) | 5.92 (2.01)

24. Secondary Outcome: Visual Analog Scale (VAS) Question: Calm
Description: Visual Analog Scale (VAS) question: Calm. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 74.35 (3.60) | 76.52 (3.58)
  Day 2; post-2nd scan: number analyzed (Participants) | 59 | 58
  Day 2; post-2nd scan | 73.15 (3.60) | 69.23 (3.62)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 65.65 (3.71) | 61.15 (3.71)
  Day 3; abstinence PM: number analyzed (Participants) | 53 | 54
  Day 3; abstinence PM | 58.92 (3.73) | 52.44 (3.71)
  Day 4; abstinence AM: number analyzed (Participants) | 54 | 53
  Day 4; abstinence AM | 60.23 (3.71) | 57.97 (3.73)
  Day 4; abstinence PM: number analyzed (Participants) | 54 | 51
  Day 4; abstinence PM | 65.47 (3.71) | 62.48 (3.78)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 67.60 (3.78) | 61.02 (3.65)
  Day 5; after smoking: number analyzed (Participants) | 57 | 49
  Day 5; after smoking | 69.27 (3.65) | 70.52 (3.83)

25. Secondary Outcome: Visual Analog Scale (VAS) Question: Depressed
Description: Visual Analog Scale (VAS) question: Depressed. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 3.97 (1.52) | 2.87 (1.52)
  Day 2; post-2nd scan: number analyzed (Participants) | 59 | 58
  Day 2; post-2nd scan | 4.99 (1.52) | 5.55 (1.53)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 6.43 (1.57) | 6.85 (1.57)
  Day 3; abstinence PM: number analyzed (Participants) | 53 | 54
  Day 3; abstinence PM | 4.61 (1.58) | 4.58 (1.57)
  Day 4; abstinence AM: number analyzed (Participants) | 54 | 53
  Day 4; abstinence AM | 5.51 (1.57) | 5.17 (1.58)
  Day 4; abstinence PM: number analyzed (Participants) | 54 | 51
  Day 4; abstinence PM | 5.67 (1.57) | 5.73 (1.60)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 2.64 (1.54) | 5.26 (1.60)
  Day 5; after smoking: number analyzed (Participants) | 57 | 49
  Day 5; after smoking | 2.53 (1.54) | 4.89 (1.63)

26. Secondary Outcome: Visual Analog Scale (VAS) Question: Drowsy
Description: Visual Analog Scale (VAS) question: Drowsy. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 16.63 (3.53) | 14.29 (3.51)
  Day 2; post-2nd scan: number analyzed (Participants) | 59 | 58
  Day 2; post-2nd scan | 24.25 (3.53) | 30.17 (3.55)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 17.14 (3.65) | 15.43 (3.65)
  Day 3; abstinence PM: number analyzed (Participants) | 53 | 54
  Day 3; abstinence PM | 24.71 (3.67) | 24.36 (3.65)
  Day 4; abstinence AM: number analyzed (Participants) | 54 | 53
  Day 4; abstinence AM | 19.56 (3.65) | 18.32 (3.67)
  Day 4; abstinence PM: number analyzed (Participants) | 54 | 51
  Day 4; abstinence PM | 19.84 (3.65) | 20.50 (3.72)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 23.01 (3.58) | 21.01 (3.72)
  Day 5; after smoking: number analyzed (Participants) | 57 | 49
  Day 5; after smoking | 20.45 (3.58) | 21.45 (3.78)

27. Secondary Outcome: Visual Analog Scale (VAS) Question: Anxious
Description: Visual Analog Scale (VAS) question: Anxious. Scale ranges from 0 to 100 with higher levels indicating greater intensity of symptom/feeling.
Time Frame: Day 2 (pre and post scan), day 3 (AM and PM), day 4 (AM and PM), day 5 (pre and post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 16.69 (3.30) | 15.62 (3.28)
  Day 2; post-2nd scan: number analyzed (Participants) | 59 | 58
  Day 2; post-2nd scan | 15.02 (3.30) | 12.65 (3.31)
  Day 3; abstinence AM: number analyzed (Participants) | 54 | 54
  Day 3; abstinence AM | 20.20 (3.38) | 17.38 (3.38)
  Day 3; abstinence PM: number analyzed (Participants) | 53 | 54
  Day 3; abstinence PM | 16.38 (3.40) | 20.23 (3.38)
  Day 4; abstinence AM: number analyzed (Participants) | 54 | 53
  Day 4; abstinence AM | 18.46 (3.38) | 15.08 (3.40)
  Day 4; abstinence PM: number analyzed (Participants) | 54 | 51
  Day 4; abstinence PM | 15.88 (3.38) | 15.63 (3.44)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 57 | 51
  Day 5; after scan, pre-smoking | 17.81 (3.33) | 19.05 (3.44)
  Day 5; after smoking: number analyzed (Participants) | 57 | 49
  Day 5; after smoking | 16.26 (3.33) | 15.30 (3.48)

28. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Negative Affect
Description: Positive and Negative Affect Schedule (PANAS) Negative Affect Score. Ranges from 10-50 with higher scores representing higher levels of negative affect.
Time Frame: as for outcome 3
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 1; pre-1st smoking session: number analyzed (Participants) | 57 | 62
  Day 1; pre-1st smoking session | 11.94 (0.45) | 11.43 (0.44)
  Day 1; post-1st smoking session: number analyzed (Participants) | 55 | 59
  Day 1; post-1st smoking session | 10.64 (0.46) | 10.57 (0.45)
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 11.25 (0.45) | 11.03 (0.44)
  Day 2; post-2nd scan: number analyzed (Participants) | 55 | 56
  Day 2; post-2nd scan | 11.59 (0.46) | 11.49 (0.45)
  Day 3; abstinence AM: number analyzed (Participants) | 55 | 55
  Day 3; abstinence AM | 12.31 (0.46) | 13.01 (0.46)
  Day 3; abstinence PM: number analyzed (Participants) | 56 | 56
  Day 3; abstinence PM | 13.07 (0.45) | 12.89 (0.45)
  Day 4; abstinence AM: number analyzed (Participants) | 56 | 55
  Day 4; abstinence AM | 12.51 (0.45) | 13.06 (0.46)
  Day 4; abstinence PM: number analyzed (Participants) | 56 | 53
  Day 4; abstinence PM | 12.90 (0.45) | 13.16 (0.46)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 56 | 50
  Day 5; after scan, pre-smoking | 12.55 (0.45) | 12.18 (0.47)
  Day 5; after smoking: number analyzed (Participants) | 52 | 48
  Day 5; after smoking | 11.41 (0.47) | 11.94 (0.48)

29. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Positive Affect
Description: Positive and Negative Affect Schedule (PANAS) Positive Affect Score. Ranges from 10-50 with higher scores representing higher levels of positive affect.
Time Frame: as for outcome 3
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 1; pre-1st smoking session: number analyzed (Participants) | 59 | 62
  Day 1; pre-1st smoking session | 37.10 (1.24) | 37.23 (1.23)
  Day 1; post-1st smoking session: number analyzed (Participants) | 56 | 59
  Day 1; post-1st smoking session | 35.72 (1.25) | 36.11 (1.24)
  Day 2; pre-1st scan: number analyzed (Participants) | 59 | 60
  Day 2; pre-1st scan | 36.08 (1.24) | 36.55 (1.23)
  Day 2; post-2nd scan: number analyzed (Participants) | 56 | 56
  Day 2; post-2nd scan | 33.51 (1.25) | 34.17 (1.25)
  Day 3; abstinence AM: number analyzed (Participants) | 56 | 56
  Day 3; abstinence AM | 32.57 (1.25) | 33.30 (1.25)
  Day 3; abstinence PM: number analyzed (Participants) | 56 | 56
  Day 3; abstinence PM | 32.34 (1.25) | 32.81 (1.25)
  Day 4; abstinence AM: number analyzed (Participants) | 56 | 55
  Day 4; abstinence AM | 32.56 (1.25) | 32.03 (1.25)
  Day 4; abstinence PM: number analyzed (Participants) | 56 | 53
  Day 4; abstinence PM | 33.25 (1.25) | 32.61 (1.26)
  Day 5; after scan, pre-smoking: number analyzed (Participants) | 55 | 50
  Day 5; after scan, pre-smoking | 33.45 (1.25) | 32.53 (1.27)
  Day 5; after smoking: number analyzed (Participants) | 54 | 48
  Day 5; after smoking | 33.10 (1.25) | 33.76 (1.27)

30. Secondary Outcome: Nicotine Effects Questionnaire (NEQ) Question: Feels Strength of Nicotine
Description: Nicotine Effects Questionnaire (NEQ) question: feels strength of nicotine. Score ranges from 0 to 100 with higher levels indicating feeling stronger effects of nicotine after smoking.
Time Frame: Day 1 (pre smoking session), Day 5 (post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 1; pre-1st smoking session: number analyzed (Participants) | 54 | 56
  Day 1; pre-1st smoking session | 71.45 (3.55) | 71.01 (3.51)
  Day 5; after smoking: number analyzed (Participants) | 52 | 44
  Day 5; after smoking | 74.87 (3.60) | 75.25 (3.79)

31. Secondary Outcome: Nicotine Effects Questionnaire (NEQ) Question: Feels Good Effects of Nicotine
Description: NEQ question: feels good effects of nicotine. Score ranges from 0 to 100 with higher levels indicating feeling more good effects of nicotine after smoking.
Time Frame: Day 1 (pre smoking session), Day 5 (post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 1; pre-1st smoking session: number analyzed (Participants) | 54 | 56
  Day 1; pre-1st smoking session | 67.72 (3.75) | 67.84 (3.71)
  Day 5; after smoking: number analyzed (Participants) | 52 | 44
  Day 5; after smoking | 67.84 (3.80) | 64.72 (3.99)

32. Secondary Outcome: Nicotine Effects Questionnaire (NEQ) Question: Feels Bad Effects of Nicotine
Description: Nicotine Effects Questionnaire (NEQ) question: feels bad effects of nicotine. Score ranges from 0 to 100 with higher levels indicating feeling more bad effects of nicotine after smoking.
Time Frame: Day 1 (pre smoking session), Day 5 (post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 1; pre-1st smoking session: number analyzed (Participants) | 54 | 56
  Day 1; pre-1st smoking session | 26.25 (3.91) | 25.92 (3.86)
  Day 5; after smoking: number analyzed (Participants) | 52 | 44
  Day 5; after smoking | 25.39 (3.96) | 28.70 (4.19)

33. Secondary Outcome: Nicotine Effects Questionnaire (NEQ) Question: Head Rush
Description: Nicotine Effects Questionnaire (NEQ) question: feels head rush. Score ranges from 0 to 100 with higher levels indicating feeling stronger/more intense head rush after smoking.
Time Frame: Day 1 (pre smoking session), Day 5 (post smoking session)
Population: Some data is missing due to participants missing/skipping visits or from withdrawing or being withdrawn from the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Progesterone 200 mg Capsules | Progesterone 200 mg Look-alike Capsules
Number analyzed (Participants) | 66 | 66
score on a scale
  Day 1; pre-1st smoking session: number analyzed (Participants) | 54 | 56
  Day 1; pre-1st smoking session | 30.58 (4.65) | 29.38 (4.59)
  Day 5; after smoking: number analyzed (Participants) | 52 | 44
  Day 5; after smoking | 40.23 (4.71) | 42.48 (5.01)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the duration of the study (2-3 months from first visit in phase 1 to final visit in phase 2 of crossover design)
Groups:
- Progesterone 200 mg Look-alike Capsules: This arm includes all phases when participants were received placebo (phase 1/week 1 for participants randomized to receive placebo first; phase 2/week 2 for participants randomized to receive placebo second)
- Progesterone 200 mg Capsules: This arm includes all phases when participants were received progesterone (phase 1/week 1 for participants randomized to receive progesterone first; phase 2/week 2 for participants randomized to receive progesterone second)
Arm/Group | Progesterone 200 mg Look-alike Capsules | Progesterone 200 mg Capsules
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 54/66 | 56/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone 200 mg Look-alike Capsules (N=66) | Progesterone 200 mg Capsules (N=66)
Headache (Nervous system disorders) | 16 (18) | 12 (13)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (7) | 6 (6)
Irritability (Psychiatric disorders) | 30 (39) | 27 (37)
Insomnia (Psychiatric disorders) | 8 (10) | 3 (3)
Hypersomnia (Psychiatric disorders) | 3 (3) | 5 (9)
Lightheadedness (Nervous system disorders) | 2 (2) | 1 (1)
Other adverse event (General disorders) | 47 (117) | 47 (107)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT01954966/Prot_SAP_000.pdf